CLINICAL TRIAL: NCT00028366
Title: A Randomized, Comparative Study of Lopinavir/Ritonavir Versus GW433908 and Ritonavir Versus Lopinavir/Ritonavir and GW433908 (In Combination With Tenofovir Disoproxil Fumarate and One or Two Nucleoside Reverse Transcriptase Inhibitors) in HIV-1-Infected Subjects With Virologic Treatment Failure
Brief Title: Dual Versus Triple Protease Inhibitor Combinations, Including Ritonavir, in HIV Infected People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5143; 10681 (Registry Identifier: DAIDS ES); ACTG A5143; AACTG A5143; Substudy AACTG A5147S; Substudy ACTG A5147S
Record Dates: First submitted 2001-12-27; First posted 2001-12-28 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; RNA, Viral; Reverse Transcriptase Inhibitors; Viral Load; ABT 378; tenofovir disoproxil; VX-175; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — fosamprenavir; Lopinavir; Ritonavir; Tenofovir

INTERVENTIONS:
Drug: Fosamprenavir
Drug: Lopinavir/Ritonavir
Drug: Ritonavir
Drug: Tenofovir disoproxil fumarate

SUMMARY:
Ritonavir (RTV) is a protease inhibitor (PI) commonly used to increase drug levels of other PIs in HIV drug treatment. The purpose of this study is to compare a combination of drugs which includes RTV and 2 protease inhibitors (PIs) with 2 combinations that include RTV and another PI. This study also will compare the effectiveness, safety, tolerability, and drug levels in the blood of these anti-HIV drug combinations.

DETAILED DESCRIPTION:
A substantial proportion of patients on antiretroviral therapy do not achieve sustained suppression of HIV viral load. Developing strategies to improve responses to subsequent regimens is an important objective for the management of patients with HIV infection. Increasing the potency of regimens by using a pharmacoenhancer such as RTV is of interest. RTV is used widely to increase plasma concentrations of PIs, but there is little efficacy and tolerability data about different RTV-enhanced PIs. The efficacy and tolerability of a triple PI regimen will be compared to dual PI regimens; dual PI regimens will also be compared to each other.

In Step 1, patients will be selectively randomized (based on prior exposure to the study drugs) and enrolled into 1 of 3 study arms. Patients in Arm A will receive lopinavir (LPV)/RTV in combination with TDF and 1 or 2 other NRTIs; patients in Arm B will receive fosamprenavir plus RTV in combination with TDF and 1 or 2 other NRTIs; Arm C patients were to receive LPV/RTV plus fosamprenavir in combination with TDF and 1 or 2 other NRTIs. Because interim study results indicated that mean PI levels for patients in Arm C were unacceptably low, Arm C patients will now either drop LPV/RTV and add RTV or drop fosamprenavir from their regimens.

The study will last 24 to 48 weeks. Medications and clinical assessment and blood collection will be performed at 2 weeks prior to entry, entry, and Weeks 2, 4, 8, 12, 16, 24, 32, 40, and 48. Blood samples to test for amprenavir (APV) and LPV pharmacokinetics will be collected at Weeks 12, 24, 48, and at confirmed virologic failure visits. In substudy A5147S, intensive 12-hour pharmacokinetic sampling for APV, LPV, and RTV will be conducted. The first 20-25 patients enrolled in each arm will be enrolled in the substudy 14-28 days after starting study treatment.

ELIGIBILITY:
Note: Accrual into A5143 and A5147S has been discontinued. The study originally planned to enroll 216 participants, but only 56 participants were enrolled at the time of early termination of enrollment because of interim review results.

Inclusion Criteria for Step 1

* HIV infected
* Past anti-HIV therapy consisting of at least 1 PI-containing regimen or detectable viral load, and at least 1 year total anti-HIV therapy experience
* Viral load of more than 5000 copies/ml within 60 days prior to screening while on a stable anti-HIV therapy for at least 12 weeks
* Agree to use acceptable forms of contraception

Exclusion Criteria

* More than 7 days of treatment with LPV and/or more than 7 days of treatment with APV or fosamprenavir
* HIV vaccine within 90 days of study entry
* Experimental drugs within 30 days of study entry
* Cancer chemotherapy within 30 days of study entry
* Drugs that affect the immune system within 30 days of study entry
* Certain drugs within 14 days of study entry. Patients who have used drugs that might damage the kidneys within 7 days of study entry are allowed.
* Midazolam within 7 days of study entry
* Allergic or sensitive to study drugs
* Excessive drug or alcohol use
* Serious illness requiring treatment and/or hospitalization and have not completed therapy, or are not stable on therapy for at least 14 days prior to study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann C. Collier, MD, Study Chair — University of Washington
Locations (13):
- United States (13):
  - USC CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Cooper CL, van Heeswijk RP, Gallicano K, Cameron DW. A review of low-dose ritonavir in protease inhibitor combination therapy. Clin Infect Dis. 2003 Jun 15;36(12):1585-92. doi: 10.1086/375233. Epub 2003 Jun 5. PMID 12802760
- [Background] Cvetkovic RS, Goa KL. Lopinavir/ritonavir: a review of its use in the management of HIV infection. Drugs. 2003;63(8):769-802. doi: 10.2165/00003495-200363080-00004. PMID 12662125
- [Background] Moyle GJ, Back D. Principles and practice of HIV-protease inhibitor pharmacoenhancement. HIV Med. 2001 Apr;2(2):105-13. doi: 10.1046/j.1468-1293.2001.00063.x. PMID 11737387
- [Background] Nadler J. New anti-HIV protease inhibitors provide more treatment options. AIDS Patient Care STDS. 2003 Nov;17(11):551-64. doi: 10.1089/108729103322555944. PMID 14746663
- [Background] van Heeswijk RP, Veldkamp A, Mulder JW, Meenhorst PL, Lange JM, Beijnen JH, Hoetelmans RM. Combination of protease inhibitors for the treatment of HIV-1-infected patients: a review of pharmacokinetics and clinical experience. Antivir Ther. 2001 Dec;6(4):201-29. PMID 11878403
- [Result] Kashuba AD, Tierney C, Downey GF, Acosta EP, Vergis EN, Klingman K, Mellors JW, Eshleman SH, Scott TR, Collier AC. Combining fosamprenavir with lopinavir/ritonavir substantially reduces amprenavir and lopinavir exposure: ACTG protocol A5143 results. AIDS. 2005 Jan 28;19(2):145-52. doi: 10.1097/00002030-200501280-00006. PMID 15668539